CLINICAL TRIAL: NCT01916577
Title: Autologous CD117+ Progenitor Cell Mobilization for Lung Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-0388; 11BGF-31, Project #:2565477 (Other Grant/Funding Number: Colorado State BDEG Grant #: 11BGF-31, Project #:2565477); MAMO0811-1 (Other: Sanofi)
Record Dates: First submitted 2013-07-29; First posted 2013-08-05 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: COPD; Cystic Fibrosis; Pulmonary Fibrosis
Keywords: Stem Cell Mobilization; Stem Cells; Transplantation; Autologous
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cystic Fibrosis; Pulmonary Fibrosis | interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plerixafor (Mozobil) Control Arm (Active Comparator): Plerixafor mobilization of autologous CD117 stem cells: Plerixafor will be given at 240mcg/kg subcutaneously once to 5 normal control patients (volunteers) at time zero with blood collected for flow cytometric analysis for CD117+ peripheral blood cells prior to the dose and then again 8 hours after the dose
  Interventions: Drug: Plerixafor mobilization of autologous CD117 stem cells
- Plerixafor (Mozobil) Experimental Arm (Experimental): Plerixafor mobilization of autologous CD117 stem cells: Plerixafor will be given at 240mcg/kg subcutaneously once to 5 COPD, 5 Cystic Fibrosis, and 5 Pulmonary Fibrosis patients (awaiting lung transplantation) at time zero with blood collected for flow cytometric analysis for CD117+ peripheral blood cells just prior to the dose and then again 8 hours after the dose
  Interventions: Drug: Plerixafor mobilization of autologous CD117 stem cells

INTERVENTIONS:
Drug: Plerixafor mobilization of autologous CD117 stem cells — Peripheral mobilization of autologous CD117+ stem cells from the bone marrow in patients awaiting lung transplantation versus normal controls
  Other Names: Mozobil

SUMMARY:
The purpose of this study is to determine if the drug Plerixafor (Mozobil) can lead to clinically relevant efflux of CD117+ stem cells from the bone marrow to the peripheral blood of normal controls and patients awaiting lung transplantation. The investigator's hypothesis is that Plerixafor (Mozobil) will lead to significant mobilization of CD117+ stem cells to the peripheral blood.

DETAILED DESCRIPTION:
The investigators have developed a new therapy utilizing a stem cell found in the bone marrow that is defined by cell surface expression of the protein "cluster of differentiation antigen 117" (CD117). Studies utilizing these stem cells in a mouse heart transplant model have demonstrated significantly improved survival of transplanted hearts, (as much as more than 5 times that seen with untreated heart transplants). In vitro studies in mice also show that these cells work to inhibit the immune system by inhibiting T cell activation/proliferation by both paracrine (primary) and contact-dependent (lesser) mechanisms. Importantly, these stem cells are taken from the intended transplant recipient (autologous) and since these cells are part of their own body normally (in small numbers); these cells are theoretically without risk to the patient. This is very different from other stem cell therapies, which are taken from the donor and as such put the patient at significant risk of developing potentially life-threatening immune reactions. Because the use of our own stem cells is potentially safe - the rapid study, development, and implementation of autologous CD117 stem cell (SC) therapy in human transplant patients is theoretically possible. Therefore, these cells have high impact potential for the field of tissue and organ transplantation as well as auto-immunity - to potentially improve tissue/cellular engraftment, decrease acute rejection, and/or to promote organ transplant tolerance (lack of rejection despite no concomitant immune-suppression). Prior to full clinical development (efficacy trials in humans), the next step is to develop a safe and efficacious means for obtaining relatively large quantities of these cells from potential human recipients. As bone marrow biopsy for cell capture is not without risk (especially to ill potential lung transplant recipients), the investigators propose to use Plerixafor (Mozobil), a CXC-chemokine receptor 4 (CXCR4)-inhibitor to cause efflux of bone marrow-derived CD117+ cells to the peripheral blood for capture by apheresis/positive selection. If successful, the next step will be to perform initial safety studies in human patients awaiting transplantation and normal controls (not a goal of this initial protocol however). These studies have the potential to lead to large-scale clinical efficacy trials and ultimate indication/implementation for human disease(s).

Primary Outcome Measure: The number of circulating CD117+ cells per milliliter (ml) of peripheral blood at baseline and following Plerixafor (Mozobil) treatment (change in peripheral blood CD117+ cells per ml).

Secondary Outcome Measures:

i.) The number of Plerixafor (Mozobil) related adverse events (AEs). ii.) The number of patients with Plerixafor (Mozobil) related AEs iii.) The number of Plerixafor (Mozobil) related serious adverse events (SAEs). iv.) The number of patients with Plerixafor (Mozobil) related serious adverse events (SAEs).

As listed in the package insert, the most common adverse reactions (≥10%) during hematopoietic stem cell mobilization were: diarrhea (37%), nausea (34%), fatigue (27%), injection site reaction (34%), headache (22%), arthralgia (13%), dizziness (11%), and vomiting (10%). It should be noted that the majority of these occurred in patients also undergoing apheresis.

Outcome Measure Time Frame:

Primary Outcome Measure Time Frame: At baseline and at 8 hours post-Plerixafor (Mozobil) treatment

Secondary Outcome Measures Time Frame:

i.): Continuously for the first 30 minutes post-Plerixafor (Mozobil) treatment, at 1 week post-Plerixafor (Mozobil) treatment, and up to 1 year post treatment.

ii.): For the first 30 minutes post administration, at 1 week post-Plerixafor (Mozobil) treatment and up to 1 year post treatment, at 1 week post-Plerixafor (Mozobil) treatment, and up to 1 year post treatment.

iii.): For the first 30 minutes post administration, at 1 week post-Plerixafor (Mozobil) treatment and up to 1 year post treatment, at 1 week post-Plerixafor (Mozobil) treatment, and up to 1 year post treatment.

iv.): For the first 30 minutes post administration, at 1 week post-Plerixafor (Mozobil) treatment and up to 1 year post treatment, at 1 week post-Plerixafor (Mozobil) treatment, and up to 1 year post treatment.

Primary Study Goals:

To determine whether Plerixafor (Mozobil) will mobilize CD117+ progenitor cells from the bone marrow in patients with chronic lung diseases on the lung transplant waiting list (versus normal controls). We will compare baseline counts of CD117+ cells with cell counts 8 hrs after Plerixafor to determine the efficacy of mobilization.

The primary results will be used to determine the number of rounds of apheresis that may be required to isolate sufficient cells for reinfusion at later timepoints in a future study.

Significance:

If the investigators can mobilize a sufficient number of autologous CD117+ cells, they will eventually re-infuse them at the time of transplant to determine whether we can abrogate acute rejection following human lung transplantation (future study). The investigators believe these are safer than allogeneic stem cells as there is no risk for graft versus host disease (GVHD) with autologous cells.

Hypothesis:

These experiments should demonstrate the effectiveness of CD117+ stem cell mobilization from the bone marrow to the peripheral blood (PB) via CXCR4 antagonism (Plerixafor) and whether end-stage lung disease affects the ability to mobilize stem cells. Additionally, these results will be used to mathematically extrapolate approximately how many rounds of peripheral blood apheresis will be required to attain adequate stem cell numbers for clinical infusion (10e7) for a future study.

Methods:

Experiments will involve taking blood from consented patients awaiting lung transplantation (as well as normal controls) prior to Plerixafor (Mozobil) treatment (240mcg/kg subcutaneously) and then 8 hours after treatment as in Table 1.

TABLE 1:

Patient Category PB baseline analysis Plerixafor (Mozobil) Rx PB analysis 8hrs post-Rx

Awaiting Tx (n=15, 5 chronic obstructive pulmonary disease (COPD), 5 Cystic Fibrosis (CF), and 5 Pulmonary Fibrosis (PF)) CD117 isolation/analysis by Flow Cytometry Yes - 240 mcg/kg CD117+ stem cell isolation/analysis by Flow Cytometry

Normal Control (n=5) CD117 isolation/analysis by Flow Cytometry Yes - 240mcg/kg CD117+ stem cell isolation/analysis by Flow Cytometry

ELIGIBILITY:
Inclusion Criteria:

* Patients on the Univ. of Colorado Lung Transplant Waiting List Age 18 to 70 years old Ability to sign and understand informed consent
* Patients 18 years or older up to age 70 on the University of Colorado Lung Transplant Waiting List and normal control subjects will be eligible for enrollment. Patients will include those with Chronic Obstructive Lung Disease, Pulmonary Fibrosis and Cystic Fibrosis

Normal control subjects = 5

Lung Transplant waitlist patients = 15 (5 each with COPD, PF or CF to determine whether disease affects mobilization potential)

Exclusion Criteria:

* Subject has already undergone lung transplantation.
* Subject has a known or suspected allergy to Plerixafor.
* Women of child-bearing age who are unwilling to use appropriate birth control to prevent becoming pregnant.
* Subjects who have received an investigational agent or device within 30 days of administration of the study agent. For the purposes of this trial, an investigational agent or device is any which is implemented under an Investigational New Drug Application (IND).
* Subjects with a history of Hepatitis B or C.
* Subjects with significant anemia (HCT < 35),thrombocytopenia (Plt count <100,000/cc), leukocytosis (WBC > 12,000/cc), or leucopenia (WBC < 5,000/cc).
* Subjects with splenomegaly.
* Subjects unable to comply with all protocol requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-08; Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The number of circulating CD117+ cells per milliliter (ml) of peripheral blood at baseline and following Plerixafor (Mozobil) treatment (change in peripheral blood CD117+ cells per ml). | At baseline and at 8 hours post-Plerixafor (Mozobil) treatment

SECONDARY OUTCOMES:
The number of Plerixafor (Mozobil) related adverse events (AEs) | For 30 minutes after administration, at 1 week post-Plerixafor (Mozobil) treatment and up to 1 year post treatment.
The number of patients with Plerixafor (Mozobil) related adverse events | For the first 30 minutes post administration, at 1 week post-Plerixafor (Mozobil) treatment and up to 1 year post treatment
The number of Plerixafor (Mozobil) related serious adverse events (SAEs). | For the first 30 minutes post administration, at 1 week post-Plerixafor (Mozobil) treatment and up to 1 year post treatment
The number of patients with Plerixafor (Mozobil) related serious adverse events (SAEs) | For the first 30 minutes post administration, at 1 week post-Plerixafor (Mozobil) treatment and up to 1 year post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Todd Grazia, M.D., Principal Investigator — The University of Colorado Denver - Anschutz Medical Campus
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

REFERENCES:
- [Background] Blum A, Childs RW, Smith A, Patibandla S, Zalos G, Samsel L, McCoy JP, Calandra G, Csako G, Cannon RO 3rd. Targeted antagonism of CXCR4 mobilizes progenitor cells under investigation for cardiovascular disease. Cytotherapy. 2009;11(8):1016-9. doi: 10.3109/14653240903131640. PMID 19929465
- [Background] Bonig H, Chudziak D, Priestley G, Papayannopoulou T. Insights into the biology of mobilized hematopoietic stem/progenitor cells through innovative treatment schedules of the CXCR4 antagonist AMD3100. Exp Hematol. 2009 Mar;37(3):402-15.e1. doi: 10.1016/j.exphem.2008.10.017. Epub 2009 Jan 20. PMID 19157683
- [Background] D'Addio A, Curti A, Worel N, Douglas K, Motta MR, Rizzi S, Dan E, Taioli S, Giudice V, Agis H, Kopetzky G, Soutar R, Casadei B, Baccarani M, Lemoli RM. The addition of plerixafor is safe and allows adequate PBSC collection in multiple myeloma and lymphoma patients poor mobilizers after chemotherapy and G-CSF. Bone Marrow Transplant. 2011 Mar;46(3):356-63. doi: 10.1038/bmt.2010.128. Epub 2010 May 31. PMID 20577218